CLINICAL TRIAL: NCT01853111
Title: Biomarker-guided Withdrawal of Immunosuppression in Recipients of Vascularized Composite Tissue Transplants
Brief Title: Withdrawal of Immunosuppression in Recipients of Face and Extremity Transplants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Bodhan Pomahac, Director, Plastic Surgery Transplantation, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012P001539
Record Dates: First submitted 2013-05-10; First posted 2013-05-14 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Vascularized Composite Allotransplantation
MeSH Terms: interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interleukin 2 (Experimental): Subjects who receive a tolerogenic drug protocol
  Interventions: Biological: Interleukin-2

INTERVENTIONS:
Biological: Interleukin-2
  Other Names: Aldesleukin, proleukin

SUMMARY:
Many patients suffer from devastating injuries to vascularized composite tissues. Vascularized composite tissues are blocs of functional tissue that can contain multiple tissue types such as bone, muscle, nerves, blood vessels, tendons, ligaments, and others. Examples of patients with severe vascularized composite tissue defects include limb amputees, patients with third-degree burns to the face or extremities, soldiers with improvised-explosive-device blast injuries to the face, and others. These patients cannot be helped satisfactorily with conventional reconstructive surgery; however, recently vascularized composite allotransplantation (VCA) such as transplantation of faces and limbs became available to this patients. Unfortunately, at this juncture, patients who receive VCA must submit to life-long regime of immunosuppressant drugs with serious side effects such as infection, renal toxicity and cancer. Immune tolerance is the absence of a destructive immune response from the recipient's body to the transplant, while otherwise maintaining sufficient immune function to fight infections and other threats. Transplant recipients with immune tolerance do not need to take immunosuppression drugs. The investigators believe that they can achieve immune tolerance in recipients of face and limb transplants.

ELIGIBILITY:
Inclusion Criteria:

* adults who have received VCA transplants at Brigham and Women's Hospital
* no less than 3 months elapsed since VCA transplant,
* on steroid-free immune dual immunosuppression with tacrolimus (6-8 ng/ml trough levels) and mycophenolate mofetil,
* no current concerns of rejection

Exclusion Criteria:

* recent (<3 months) episodes of rejection,
* active bacterial or viral infection,
* malignancy,
* non-healing wounds
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Complete cessation of immune suppression without evidence of rejection for more than 6 months. | 6 -24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Pomahac, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States